CLINICAL TRIAL: NCT00941824
Title: Pharmacokinetic Evaluation of an Intensified and Decreasing Dosing Regimen of Mycophenolate Sodium in Combination With Tacrolimus During the First 3 Months Post Kidney Transplant (the myFORTic Study)
Brief Title: Pharmacokinetic Evaluation of an Intensified and Decreasing Dosing Regimen of Mycophenolate Sodium in Combination With Tacrolimus Post Kidney Transplant: The Myfortic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément Caillaux,, CHU SAINT-ETIENNE
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0808100; 2009-010710-29
Record Dates: First submitted 2009-07-09; First posted 2009-07-20 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Kidney Transplantation
Keywords: pharmacokinetic; mycophénolate acid; kidney transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: mycophénolate acid — * Day 0 to Day 7, 720 mg twice daily
  * Day 8 to Day 30, 540 mg twice daily
  * Day 30 to Day 90, 360 mg twice daily

SUMMARY:
Mycophenolate acid (MPA) has been developed and approved in combination with cyclosporine and has been used in kidney transplantation for more than a decade. At present, combination of tacrolimus and mycophenolate acid tends to be considered as the standard of care for maintenance immunosuppression in kidney transplantation. Mainly due to a different effect on the entero-hepatic recycling pathway, cyclosporine and tacrolimus differently interfere with MPA clearance. When used with tacrolimus, MPA dosage has thus to be adjusted and cannot be extrapolated from what is recommended for a cyclosporine-based treatment. However, there is currently no clear guideline for MPA dosing when this drug is used in combination with tacrolimus. This is potentially detrimental for patients since under-or overexposure of MPA has been clinically linked to the outcome of transplantation.

The purpose of this study is to pharmacologically validate an original MPA dosing regimen in combination with tacrolimus within the three months post-kidney transplant. This regimen consists in an intensified dosing of mycophenolate sodium during the earliest period of transplantation in order to rapidly reach the appropriate MPA blood exposure followed by a gradual decrease in dose in order to prevent MPA overexposure.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Renal transplant from a dead or alive donor.
* Patients treated by initial quadritherapy with basiliximab, tacrolimus, steroid et mycophenolate sodic
* ΒHCG pregnancy test negative at the initiation of Myfortic ®
* Effective contraception during treatment and up to 6 weeks after treatment with Myfortic ®

Exclusion Criteria:

* Patient at high risk of rejection of a transplant
* IMC > ou = 30
* Platelets < 75000 / mm3 and/or neutrophils < 1500 / mm3 and/or leukocytes < 2500/ mm3 and/or hemoglobin < 6 g/dL.
* Patient requiring a anti-CMV prophylaxis by valganciclovir.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC0 - 12 hours) of the MPA and its métabolites MPAG and Ac-MPAG | at Day 2, Day 7, Day 15, Month 1, Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Mariat, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Departement of Nephrology CHU Saint-Etienne, Saint-Etienne, France